CLINICAL TRIAL: NCT06873568
Title: A Post-market Study Evaluating Clinical and Safety Outcomes of Unipolar Hemiarthroplasty Using Cephalic Femoral Heads in Subjects with Hip Fracture
Brief Title: Cephalic Femoral Heads Follow Up
Status: Not yet recruiting | Type: Observational
Sponsor: Limacorporate S.p.a (Industry)
Responsible Party: Sponsor
Other Study IDs: H-45
Record Dates: First submitted 2025-03-07; First posted 2025-03-12 (Actual); Last update posted 2025-03-18 (Actual); Status verified 2025-03

CONDITIONS: Hip Arthroplasty Replacement; Femoral Fractures
Keywords: femoral head; Partial hip arthroplasty
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Patients who underwent hip arthroplasty with cephalic femoral heads from 1at January 2023 onwards.: The study population for this clinical investigation includes subjects who suffered from a traumatic proximal femur fracture and underwent a Unipolar hemiarthroplasty with Cephalic femoral head from January 1st, 2023, onwards. Due to the characteristics of patients who underwent this type of surgery, it is expected that a considerable number of eligible patients would be in the elderly age.

SUMMARY:
Study design: monocentric, retrospective, observational and post-market clinical study.

Purpose: To demonstrate the safety and performance of cephalic femoral heads. The eligible study population is represented by the entire population that underwent a hip replacement with cephalic femoral heads from 1st January 2023 onwards at the site in accordance with the indication for use of the product.

DETAILED DESCRIPTION:
The study is aiming to demoranstrate safety and performance of cephalic femoral heads and will do it by considering the rate of revision of any prosthesis component and dislocation, by x-ray evaluation, by patient reported outcomes and walking/residential status. Patients are followed for 2 years after hemiarthroplasty and data are collected at 6 timepoints (pre-operative, intra-operative, at discharge, 4-months follow up, 12 months follow up and 24 months follow up).

ELIGIBILITY:
Inclusion Criteria:

* Displaced intracapsular hip fracture (Garden III-IV).
* Subjects underwent a Unipolar Hemiarthroplasty with a Cephalic femoral head as per their Indication For Use from January 1st, 2023, onwards.
* No concurrent joint disease at the time of the surgery.
* Absence of severe cognitive dysfunction demonstrated by 3 or more correct answers on the Pfeiffer test.
* Ability to ambulate independently with or without walking aids before surgery.
* Subject willingness to participate.

Exclusion Criteria:

* Undisplaced or minimally displaced intracapsular hip fracture (Garden I-II).
* Any Cephalic femoral head contraindication for use as reported in the current Instruction For Use.
* Pathological fracture secondary to malignant disease.
* Subjects with rheumatoid arthritis or symptomatic osteoarthritis.
* Previous treatment to the same hip for a fracture at the time of the surgery.
* Subjects who were deemed unsuitable for the surgical procedures by the anesthesiologist.
* Severe cognitive dysfunction or cognitive impairment demonstrated by 2 or less correct answers on the Pfeiffer test.
* Unable to walk before surgery (e.g., wheelchair or bed-ridden subjects).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent partial hip arthroplasty with cephalic femoral heads from 1st January 2023 onwards
Sampling Method: Probability Sample
Enrollment: 47 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the revision rate of Cephalic femoral heads for any reason at 24 months after Unipolar Hemiarthroplasty. | From intraoperative to 24months follow up visit

SECONDARY OUTCOMES:
Evaluation of the dislocation rate (including close reduction) in subjects with Cephalic femoral heads from intra-operative to 24 months after Unipolar Hemiarthroplasty. | From intraoperative to 24months follow up visit
Evaluation of the revision incidence of any hip component for any reason from intra-operative to 24 months after Unipolar Hemiarthroplasty. | From intraoperative to 24months follow up visit
Evaluation of acetabular erosion (according to Baker classification) in subjects with Cephalic femoral heads at 12 months after Unipolar Hemiarthroplasty. | 12 months follow up visit
  Baker classification is graded from 0 to 3, where 3 is the worst case. Grade 0: no erosion Grade 1: narrowing the arthicular cartilage, no erosion Grade 2: acetabular erosion and early migration Grade 3: protrusion acetabuli
Assessment of Harris Hip Score (HHS) at 24 months after Unipolar Hemiarthroplasty with Cephalic femoral heads. | 24 months follow up visit
  The Harris Hip Score goes from 0 to 100, which is the best result.
Assessment of Oxford Hip Score (OHS) completed by subjects with Cephalic femoral heads at 24 months after Unipolar Hemiarthroplasty. | 24 months follow up visit
  The Oxford Hip Score goes from 0 to 48, with 48 being the best outcome
Assessment of Pain Likert-scale in subjects with Cephalic femoral heads at 24 months after Unipolar Hemiarthroplasty. | 24 months follow up visit
  The pain Likert-scale is a 6-point scale:
  * severe and spontaneous
  * severe when walking
  * tollerable
  * occurs after activity
  * light intermittent
  * no pain
Comparison between pre-operative and 4-month walking ability. | Performed at preoperative visit to 4months follow up visit
  Functional evaluation
Comparison between pre-operative and 4-month residential status. | Performed at preoperative visit and 4months follow up visit
  Daily habit

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital J.A. Reimana, Prešov, Slovakia